CLINICAL TRIAL: NCT01601691
Title: Protection of Rectum From High Radiation Doses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Markku Vaarala, MD, PhD, MD, PhD, University of Oulu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 241/2011
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; brachytherapy; spacer; side effect
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spacer (Experimental): Subjects with spacer injection
  Interventions: Device: DuraSeal

INTERVENTIONS:
Device: DuraSeal — Single dose of DuraSeal product with DuraSeal components diluted 1:1 in sterile saline injected between rectum and prostate

SUMMARY:
The purpose of this study is to evaluate the usefulness of diluted DuraSeal product as a spacer between prostate and rectum in prostate cancer low dose brachytherapy.

DETAILED DESCRIPTION:
Radiation therapy for prostate cancer leads to inappropriate radiation dose to the rectum wall leading rectum adverse effects in long term for some patients. A resorbable spaces between prostate and rectum could decrease the incidence of these side effect. In this trial, men with prostate cancer with intention to curative treatment by low dose brachytherapy will be recruited. Diluted DuraSeal will be applied between rectum and prostate at the end of the brachytherapy seed implantation procedure. After the implantation of the brachytherapy seeds, a needle is placed between rectum and prostate through perineal skin under transrectal ultrasound guidance. The proper position of the needle is confirmed by the injection of 10-15 ml sterile saline solution. After that, DuraSeal components are diluted in 1:1 with sterile saline and 6-10 ml of this diluted product will be injected using DuraSeal applicator. The resolution of the spacer will be followed by repeated plain computer tomography (CT) of pelvis performed a day before operation, a day after the operation, 4 weeks after the operation and 8 weeks after the operation. In addition, magnetic resonance imaging of pelvis performed 8 to 16 weeks after the operation. The space created between prostate and rectum will be documented by plain CT and magnetic resonance imaging. Rectum radiation dose will be calculated based on these scans. Time to DuraSeal resolution will be evaluated from the scans. Possible side effects will be collected by subject interviews during follow-up visits at 4, 8 and 12 weeks after the operation.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer patients with planned low dose brachytherapy for the treatment of prostate cancer

Exclusion Criteria:

* not willing to participate this study

Ages: 50 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markku Vaarala, MD, PhD, Principal Investigator — Oulu Univeristy Hospital; Merja Korpela, MD, Study Chair — Oulu University Hospital; Vesa-Pekka Heikkilä, FL, Study Chair — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Oulu, Finland

REFERENCES:
- [Derived] Heikkila VP, Karna A, Vaarala MH. DuraSeal as a spacer to reduce rectal doses in low-dose rate brachytherapy for prostate cancer. Radiother Oncol. 2014 Aug;112(2):233-6. doi: 10.1016/j.radonc.2014.08.012. Epub 2014 Sep 4. PMID 25201125

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spacer
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Spacer
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: year] | 66 [58 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Finland | 10

OUTCOME MEASURES:

1. Primary Outcome: Spacer Volume Half Life
Description: Time to spacer resolution will be measured based on the distance between rectum wall and prostate on CT scans before operation and on defined time frame. In addition, magnetic resonance imaging of pelvis will be performed 8 to 16 weeks after the operation in order to confirm the extent of spacer. Spacer volume half life is reported.
Time Frame: 1 day, 4 weeks, 8 weeks, up-to 16 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Spacer
Number analyzed (Participants) | 10
days | 47 (12)

2. Secondary Outcome: Side Effects
Description: Possible side effects will be collected by subject interview and physical examination on specified time frame.
Time Frame: 1 day, 4 weeks, 8 weeks, 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Rectum Radiation Dose
Description: Rectum dose will be calculated based on CT scans after brachytherapy.
Time Frame: 1 day, 4 weeks, 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Spacer
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spacer (N=10)
sensation of pressure in rectum (Gastrointestinal disorders) | 1 (1)
sudden need for defecation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No